CLINICAL TRIAL: NCT06705556
Title: Effects of Pre and Post Operative Active Cycle of Breathing Technique as Add on to Routine Chest Physical Therapy on Respiratory Parameters in Coronary Artery Bypass Graft Patients
Brief Title: Effect of Active Cycle of Breathing Technique as Add on to Routine Chest Physical Therapy on Respiratory Parameters in Coronary Artery Bypass Graft Patients
Acronym: CABG ACBT ABG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sadaf Bukhari (Other)
Responsible Party: Sponsor-Investigator, Sadaf Bukhari, Principal investigator, University of Faisalabad
Organization: University of Faisalabad (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Tuf/IRB/292/24
Record Dates: First submitted 2024-11-18; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Bypass Graft
MeSH Terms: interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study was single, and assessor blinded. Participants were masked about other groups, but they were knowing what treatment they were receiving. Principal investigator was also not masked or blinded because investigator was applying the techniques on participants of both groups. So participant and principal investigator cannot be blinded. Only assessor was blind and was taken outcome measures without knowing the problem and treatment techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group:
  The intervention group (n=36) was instructed to perform the ACBT with routine chest physical therapy pre and postoperatively. The preoperative chest physical therapy was conducted 3 days before surgery and the postoperative CPT, including ACBT, was performed 3 times in the ICU for up to 5 days after surgery.
  Preoperative routine chest physical therapy sessions were followed as:
  * Incentive spirometer, 3 sessions per day, 10 repetitions
  * Percussions, 3 sessions per day, 20 repetitions
  * 3-minutes walking, 2 sessions per day
  * ACBT, 3 sessions per day
  The preoperative chest physiotherapy treatment plan was continued after CABG surgery. In addition to these, the following were included postoperatively:
  * Nebulization, 3 sessions per day
  * 3 minutes of walking, 2 sessions per day
  * ACBT, 3 sessions per day
  Interventions: Procedure: Active cycle of breathing technique, incentive spirometer, percussion, 3-minute of walking
- The control group (Experimental): The control group:
  The routine Chest physical therapy was performed 3 days before surgery at the preoperative bay and 5 days after surgery in the ICU with 3 sessions each day.
  Preoperative chest physical therapy sessions were followed as:
  * Incentive spirometer, 3 sessions per day, 10 repetitions.
  * Percussions, 3 sessions per day, 20 repetitions.
  * 3-minutes walking, 2 sessions per day The preoperative chest physiotherapy treatment plan was continued after CABG surgery. In addition to these, the following were included postoperatively:
  * Nebulization, 3 sessions per day
  * 3-minutes walking, 2 sessions per day
  Interventions: Procedure: incentive spirometer, percussion, 3-minute of walking

INTERVENTIONS:
Procedure: Active cycle of breathing technique, incentive spirometer, percussion, 3-minute of walking — The intervention group:
  patients were asked to perform Active cycle of breathing technique as add on to routine chest physical therapy such as Incentive spirometer, percussion, 3-minute of walking 3 days before surgery and five days postoperative.
  * Incentive spirometry, 3 sessions per day, 10 repetitions
  * Percussions, 3 sessions per day, 20 repetitions
  * 3-minutes walking, 2 sessions per day
  * ACBT, 3 sessions per day the following were included postoperatively:
  * Nebulization, 3 sessions per day
  * ACBT, 3 sessions per day
  Arms: The intervention group
Procedure: incentive spirometer, percussion, 3-minute of walking — The control group The routine CPT was performed 3 days before surgery at the preoperative bay and 5 days after surgery in the ICU with 3 sessions each day.
  Preoperative chest physical therapy sessions were followed as:
  * Incentive spirometry, 3 sessions per day, 10 repetitions.
  * Percussions, 3 sessions per day, 20 repetitions.
  * 3-minutes walking, 2 sessions per day The preoperative chest physiotherapy treatment plan was continued after CABG surgery. In addition to these, the following were included postoperatively:
  * Nebulization, 3 sessions per day
  * 3-minutes walking, 2 sessions per day
  Arms: The control group

SUMMARY:
A controlled trial was conducted to determine the effect of the active cycle of breathing technique (ACBT) in improving respiratory parameters after coronary artery bypass graft surgery. The main aim of this study was to determine the effects of pre and postoperative active cycle of breathing technique (ACBT) in coronary artery disease patients undergoing coronary artery bypass graft surgery in improving respiratory parameters such as arterial blood gas (ABG), oxygen saturation (SpO2) and respiratory rate. The intervention group performed an active cycle of breathing technique with routine chest physical therapy while the control group performed routine chest physical therapy. Arterial blood gas (ABG), oxygen saturation (SpO2), and respiratory rate were measured at baseline and five days after surgery, every 2 hours on postoperative days 1, 2, and 3 and 4 hours on days 4 and 5.

Participants in the intervention group performed preoperative routine chest physical therapy sessions were followed as:

* Incentive spirometry, 3 sessions per day, 10 repetitions
* Percussions, 3 sessions per day, 20 repetitions
* 3-minutes walking, 2 sessions per day
* ACBT, 3 sessions per day

The preoperative chest physiotherapy treatment plan was continued after CABG surgery. In addition to these, the following were included postoperatively:

* Nebulization, 3 sessions per day
* 3 minutes of walking, 2 sessions per day
* ACBT, 3 sessions per day While participants in the control group performed the same pre and postoperative sessions except ACBT.

DETAILED DESCRIPTION:
This single-blinded randomized controlled trial was conducted at the Faisalabad Institute of Cardiology, Faisalabad, Pakistan, to assess the effects the Active Cycle of Breathing Technique (ACBT) as add on to routine chest physical therapy in the preoperative care of coronary artery bypass graft (CABG) patients. The primary aim was to evaluate ACBT's impact on minimizing postoperative respiratory complications. A secondary aim was to educate patients in the preoperative period to reduce surgery-related stress and support respiratory drive.

Patients with coronary artery disease are generally advised bed rest to manage shortness of breath. However, CABG is an invasive procedure that involves the placement of an endotracheal tube, raising infection risks and leading to weakened respiratory muscles due to ventilation effects. Post-surgery, patients often experience reduced lung volumes and altered arterial blood gases. Adding ACBT to chest physical therapy in the preoperative period is intended to improve ventilation and arterial blood gas levels postoperatively.

The study involved 72 male and female patients, aged 30 to 65, with double or triple-vessel coronary disease and a 10 to 15-year disease history, scheduled for CABG. Screening was performed using a custom questionnaire based on inclusion and exclusion criteria, and non-probability purposive sampling was used to select participants. Patients were randomly assigned to either the intervention or control group using the lottery method. The intervention group received ACBT alongside routine chest physical therapy, while the control group received only standard chest physical therapy, both pre- and postoperatively. Patient confidentiality was maintained through informed consent.

Key study parameters included arterial blood gas (ABG) levels, oxygen saturation (SpO2), and respiratory rate, with ABG samples taken from the brachial and radial arteries and analyzed via an ABG analyzer. SpO2 was measured using a pulse oximeter, and respiratory rate was recorded on a cardiac monitor.

ELIGIBILITY:
Inclusion Criteria:

* Elective coronary artery bypass graft patients
* The study included both male and female
* 30 to 65 years old patients were included in this study
* Adults with stable coronary artery disease for the last 15 years

Exclusion Criteria:

* Patient with unstable vitals
* Preoperative pulmonary dysfunction
* COPD or Emphysema
* Asthma and Severe atelectasis
* Renal disorders
* Connected to the ventilator for more than 48 hours

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Arterial blood gas | ABG test was conducted once preoperative for both groups and after surgery every 2 hours on postoperative days 1, 2, and 3, and every 4 hours on days 4 and 5.
  Arterial Blood Gas (ABG) is a critical test used to evaluate a patient's acid-base balance, oxygenation, and ventilation status by measuring the levels of oxygen (O₂), carbon dioxide (CO₂), and bicarbonate (HCO₃-) in arterial blood.

SECONDARY OUTCOMES:
oxygen saturation (SpO₂) | SpO₂ was measured once preoperative for both groups and after surgery every 2 hours on postoperative days 1, 2, and 3, and every 4 hours on days 4 and 5.
  SpO₂ (Oxygen Saturation) is a measurement that estimates the percentage of oxygen-saturated hemoglobin in the blood. SpO₂ monitoring is vital in clinical settings, especially for patients with respiratory or cardiac conditions, during and after surgery.
Respiratory rate | Respiratory rate was measured once preoperative for both groups and after surgery every 2 hours on postoperative days 1, 2, and 3, and every 4 hours on days 4 and 5.
  Respiratory rate (RR) refers to the number of breaths a person takes per minute. It is a key vital sign used to assess breathing and overall respiratory function.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - The University of Faisalabad, Faisalabad, Punjab Province
  - Dr Sana Ashraf, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No